CLINICAL TRIAL: NCT01002339
Title: Optimum Immunosuppression in Renal Transplant Recipients at High Risk of Developing New Onset Diabetes After Transplantation: A Multicenter, Prospective, Controlled and Randomized Trial.
Brief Title: Optimum Immunosuppression in Renal Transplant Recipients.New Onset Diabetes After Transplantation
Acronym: 01-DMPT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated: higher rate of acute rejection in the Cyclosporin A group
Sponsor: Armando Torres Ramírez (Other)
Responsible Party: Sponsor-Investigator, Armando Torres Ramírez, PhD, Fundación Canaria Rafael Clavijo para la Investigación Biomédica
Organization: Fundación Canaria Rafael Clavijo para la Investigación Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FundacionRC
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Adult-Onset
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tacrolimus; Basiliximab; Prednisone; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tacrolimus with rapid steroid withdrawal (Experimental): Basiliximab induction. Tacrolimus plus Mycophenolate mofetil (MMF), and corticosteroids with rapid withdrawal after one week.
  Interventions: Drug: Tacrolimus with rapid steroid withdrawal
- Tacrolimus with steroids minimization (Active Comparator): Basiliximab induction.Tacrolimus plus Mycophenolate mofetil (MMF) and low-dose corticosteroids for 6 months with subsequent removal
  Interventions: Drug: Tacrolimus with steroids minimization
- CsA with steroid minimization (Experimental): Basiliximab induction. Ciclosporin A (CsA) plus Mycophenolate mofetil (MMF) and low-dose corticosteroids for 6 months with subsequent removal
  Interventions: Drug: CsA with steroid minimization

INTERVENTIONS:
Drug: Tacrolimus with rapid steroid withdrawal — * Basiliximab induction (4 mg i.v., days 0 and 4).
  * Corticosteroids: 0.5 gr of i.v. Methylprednisolone (MP) intraoperatively and 125 mg on the first day, followed by oral doses of prednisone rapidly tapered from 30 mg/day to complete discontinuation by postoperative day 7.
  * Tacrolimus: 0.15 mg/Kg/day to achieve target trough levels of 8-12 ng/ml for the first month and then 5-8 ng/ml.
  * Mycophenolate mofetil 1 gr b.i.d. for the first month and then 500 mg b.i.d.
  Other Names: Simulect; Dacortin; Prograf/Advagraf; Cellcept/Myfortic.
  Arms: Tacrolimus with rapid steroid withdrawal
Drug: Tacrolimus with steroids minimization — * Basiliximab induction (4 mg i.v., days 0 an 4)
  * Corticosteroids: 0.5 gr of i.v. MP intraoperatively and 60 mg on the first day, followed by oral doses of prednisone starting with 0.3 mg/Kg/day, and gradual weekly tapering to complete discontinuation over 6 months.
  * Tacrolimus 0.15 mg/Kg/day to achieve target trough levels of 8-12 ng/ml for the first month and then 5-8 ng/ml.
  * Mycophenolate mofetil 1 gr b.i.d. for the first month and then 500 mg b.i.d.
  Other Names: Simulect; Dacortin; Prograf/Advagraf; Cellcept/Myfortic.
  Arms: Tacrolimus with steroids minimization
Drug: CsA with steroid minimization — * Basiliximab induction (4 mg i.v., days 0 an 4)
  * Corticosteroids: 0.5 gr of i.v. MP intraoperatively and 60 mg on the first day, followed by oral doses of prednisone starting with 0.3 mg/Kg/day, and gradual weekly tapering to complete discontinuation over 6 months.
  * CsA 5 mg/Kg/day to achieve target trough of 150-200 ng/ml the first month and then 100-150 ng/ml.
  * Mycophenolate mofetil 1 gr b.i.d
  Other Names: Simulect; Dacortin; Sandimmun Neoral; Cellcept/Myfortic.
  Arms: CsA with steroid minimization

SUMMARY:
New onset diabetes after renal transplantation (NODAT) is a common and severe complication negatively influencing graft and patient survival. Cyclosporine (CsA) and Tacrolimus are the basis of modern immunosuppression. Tacrolimus is superior to CsA in terms of acute rejection and graft function. However, Tacrolimus increases 2 times the risk of NODAT as compared to CsA.

DETAILED DESCRIPTION:
New onset diabetes after renal transplantation (NODAT) is a common and severe complication negatively influencing graft and patient survival. CsA and Tacrolimus are the basis of modern immunosuppression. Tacrolimus is superior to CsA in terms of acute rejection and graft function. However, increases 2 times the risk of NODAT as compared to CsA. Objectives: a) To compare the incidence of NODAT and glucose intolerance with 3 different regimes: Tacrolimus with rapid steroid withdrawal; Tacrolimus with steroids minimization; and CsA with steroid minimization; b) To compare acute rejection rate, renal function and graft and patient survival between different regimes; and c) to investigate the influence of different regimes on subclinical atheromatosis. A total of 210 patients will be randomized. The primary efficacy variable will be NODAT or glucose intolerance at 1 year; secondary efficacy variables will be acute rejection, renal function, and changes of carotid intima-media thickness over time.

ELIGIBILITY:
Inclusion Criteria:

* Primary renal transplant recipients with end stage renal disease
* No prior history of diabetes mellitus before transplant
* Absence of Immunologic risk defined by the investigator criterion and Panel Reactive Antibody (PRA) < 50%
* Absence of severe infection and hepatitis C or B infection
* Efficient contraception in women during the study

Additionally must meet one of these "Metabolic Criteria

* Recipient age >or =60 or
* Recipient age between 45 and 59 years and at least one of the following metabolic criteria: Prior to transplantation Triglycerides (TGS) >200mg/dl or the combination of a body mass index (BMI)> 27 and Triglycerides>150 mg/dl or the combination of HDL-cholesterol<40 mg/dl for men or <50 mg/dl for women and Triglycerides >150 mg/dl.

Exclusion Criteria:

* Patients with type I or II diabetes prior to transplantation defined by the American Diabetes Association (ADA) criteria
* Recipient age under 45
* Patients receiving a second renal transplant
* Patients with high immunological risk or PRA (panel reactive antibody level) >or =50%
* Severe infection or hepatitis C or B infection.
* Dual renal transplant or double transplant with any other organ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2010-02; Primary Completion 2014-02 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armando Torres, PhD, Study Director — Fundación Canaria para la Investigación Biomédica Rafael Clavijo
Locations (10):
- Spain (10):
  - Antonio Osuna, Granada, Andalusia
  - Domingo Hernández, Málaga, Andalusia
  - Carlos Gómez Alamillo, Santander, Cantabria
  - Juan Manuel Díaz, Barcelona, Catalonia
  - Francisco Moreso, Barcelona, Catalonia
  - Francisco Valdés, A Coruña, Galicia
  - Carmen Díaz Corte, Oviedo, Principality of Asturias
  - Armando Torres Ramírez, San Cristóbal de La Laguna, S/C de Tenerife
  - Roberto Gallego, Las Palmas de Gran Canaria
  - Luis Pallardo, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Porrini E, Gomez MD, Alvarez A, Cobo M, Gonzalez-Posada JM, Perez L, Hortal L, Garcia JJ, Dolores Checa M, Morales A, Hernandez D, Torres A. Glycated haemoglobin levels are related to chronic subclinical inflammation in renal transplant recipients without pre-existing or new onset diabetes. Nephrol Dial Transplant. 2007 Jul;22(7):1994-9. doi: 10.1093/ndt/gfm067. Epub 2007 Mar 29. PMID 17395658
- [Background] Alvarez A, Fernandez J, Porrini E, Delgado P, Pitti S, Vega MJ, Gonzalez-Posada JM, Rodriguez A, Perez L, Marrero D, Luis D, Velazquez S, Hernandez D, Salido E, Torres A. Carotid atheromatosis in nondiabetic renal transplant recipients: the role of prediabetic glucose homeostasis alterations. Transplantation. 2007 Oct 15;84(7):870-5. doi: 10.1097/01.tp.0000284462.70064.ae. PMID 17984840
- [Background] Hernandez D, Miquel R, Porrini E, Fernandez A, Gonzalez-Posada JM, Hortal L, Checa MD, Rodriguez A, Garcia JJ, Rufino M, Torres A. Randomized controlled study comparing reduced calcineurin inhibitors exposure versus standard cyclosporine-based immunosuppression. Transplantation. 2007 Sep 27;84(6):706-14. doi: 10.1097/01.tp.0000282872.17024.b7. PMID 17893603
- [Background] Porrini E, Delgado P, Alvarez A, Cobo M, Perez L, Gonzalez-Posada JM, Hortal L, Gallego R, Garcia JJ, Checa M, Morales A, Salido E, Hernandez D, Torres A. The combined effect of pre-transplant triglyceride levels and the type of calcineurin inhibitor in predicting the risk of new onset diabetes after renal transplantation. Nephrol Dial Transplant. 2008 Apr;23(4):1436-41. doi: 10.1093/ndt/gfm762. Epub 2007 Nov 19. PMID 18029372
- [Background] Porrini E, Moreno JM, Osuna A, Benitez R, Lampreabe I, Diaz JM, Silva I, Dominguez R, Gonzalez-Cotorruelo J, Bayes B, Lauzurica R, Ibernon M, Moreso F, Delgado P, Torres A. Prediabetes in patients receiving tacrolimus in the first year after kidney transplantation: a prospective and multicenter study. Transplantation. 2008 Apr 27;85(8):1133-8. doi: 10.1097/TP.0b013e31816b16bd. PMID 18431233
- [Background] Bayes B, Moreso F, Benitez R, Torres A, Diaz JM, Granada ML, Lauzurica R, Pastor MC, Teixido J. [Post-transplant diabetes mellitus depending on the pre-transplant dialysis technique]. Nefrologia. 2008;28 Suppl 6:97-102. Spanish. PMID 18957019
- [Background] Porrini E, Bayes B, Diaz JM, Ibernon M, Benitez R, Dominguez R, Moreno JM, Delgado P, Lauzurica R, Silva I, Moreso F, Lampreabe I, Arias M, Osuna A, Torres A. Hyperinsulinemia and hyperfiltration in renal transplantation. Transplantation. 2009 Jan 27;87(2):274-9. doi: 10.1097/TP.0b013e318191a7d5. PMID 19155984
- [Background] Porrini EL, Diaz JM, Moreso F, Delgado Mallen PI, Silva Torres I, Ibernon M, Bayes-Genis B, Benitez-Ruiz R, Lampreabe I, Lauzurrica R, Osorio JM, Osuna A, Dominguez-Rollan R, Ruiz JC, Jimenez-Sosa A, Gonzalez-Rinne A, Marrero-Miranda D, Macia M, Garcia J, Torres A. Clinical evolution of post-transplant diabetes mellitus. Nephrol Dial Transplant. 2016 Mar;31(3):495-505. doi: 10.1093/ndt/gfv368. Epub 2015 Nov 3. PMID 26538615
- [Background] Rodriguez-Rodriguez AE, Trinanes J, Porrini E, Velazquez-Garcia S, Fumero C, Vega-Prieto MJ, Diez-Fuentes ML, Luis Lima S, Salido E, Torres A. Glucose homeostasis changes and pancreatic beta-cell proliferation after switching to cyclosporin in tacrolimus-induced diabetes mellitus. Nefrologia. 2015;35(3):264-72. doi: 10.1016/j.nefro.2015.05.007. Epub 2015 Jun 27. English, Spanish. PMID 26299169
- [Background] Rodriguez-Rodriguez AE, Trinanes J, Velazquez-Garcia S, Porrini E, Vega Prieto MJ, Diez Fuentes ML, Arevalo M, Salido Ruiz E, Torres A. The higher diabetogenic risk of tacrolimus depends on pre-existing insulin resistance. A study in obese and lean Zucker rats. Am J Transplant. 2013 Jul;13(7):1665-75. doi: 10.1111/ajt.12236. Epub 2013 May 7. PMID 23651473
- [Result] Delgado P, Diaz JM, Silva I, Osorio JM, Osuna A, Bayes B, Lauzurica R, Arellano E, Campistol JM, Dominguez R, Gomez-Alamillo C, Ibernon M, Moreso F, Benitez R, Lampreave I, Porrini E, Torres A. Unmasking glucose metabolism alterations in stable renal transplant recipients: a multicenter study. Clin J Am Soc Nephrol. 2008 May;3(3):808-13. doi: 10.2215/CJN.04921107. Epub 2008 Mar 5. PMID 18322043

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 2010
Groups:
- Tacrolimus With Rapid Steroid Withdrawal: Tacrolimus plus Mycophenolate mofetil (MMF), and corticosteroids with rapid withdrawal after one week.
  Tacrolimus with rapid steroid withdrawal: Tacrolimus 0.15 mg/Kg/day to achieve target trough levels of 8-12 ng/ml for the first month, and MMF 2 gr/day; steroids: 0.5 gr of Methylprednisolone (MP) intraoperatively and 125 mg on the first day, followed by oral doses of prednisone rapidly tapered from 30 mg/day to complete discontinuation by postoperative day 7. Basiliximab induction (4 mg, days 0 and 4).
- Tacrolimus With Steroids Minimization: Tacrolimus plus Mycophenolate mofetil (MMF) and low-dose corticosteroids for 6 months with subsequent removal
  Tacrolimus with steroids minimization: Tacrolimus 0.15 mg/Kg/day to achieve target trough levels of 8-12 ng/ml for the first month, and MMF 2 gr/day; steroids: 0.5 gr of MP intraoperatively and 60 mg day 1; followed by oral doses of prednisone and gradual tapering to complete discontinuation over 6 months. Basiliximab induction (4 mg, days 0 and 4).
- Cyclosporin A (CsA) With Steroid Minimization: CsA plus Mycophenolate mofetil (MMF) and low-dose corticosteroids for 6 months with subsequent removal
  CsA with steroid minimization: CsA 5 mg/Kg/day to achieve target trough of 150-200 ng/ml the first month, and similar pattern with MMF and steroids as group 2. Basiliximab induction (4 mg, days 0 and 4).
Period: Overall Study
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | Cyclosporin A (CsA) With Steroid Minimization
Started | 44 | 43 | 47
Completed | 44 | 42 | 42
Not Completed | 0 | 1 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Incorrect treatment assignment | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Lung cancer detected before transplant | 0 | 0 | 1
Not completed — Randomized. Not transplanted | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- CsA With Steroid Minimization: CsA plus Mycophenolate mofetil (MMF) and low-dose corticosteroids for 6 months with subsequent removal
  CsA with steroid minimization: CsA 5 mg/Kg/day to achieve target trough of 150-200 ng/ml the first month, and similar pattern with MMF and steroids as group 2. Basiliximab induction (4 mg, days 0 and 4).
- Total: Total of all reporting groups
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization | Total
Number analyzed (Participants) | 44 | 42 | 42 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (7.6) | 61.6 (7.3) | 60.2 (8.3) | 61.0 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 12 | 35
  Male | 33 | 30 | 30 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 44 | 42 | 42 | 128
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 44 | 42 | 42 | 128
Familiar history of diabetes (N) [Number; unit: participants]
  Yes | 3 | 4 | 9 | 16
  No | 35 | 29 | 30 | 94
  Not available | 6 | 9 | 3 | 18
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.95 (3.71) | 27.87 (3.72) | 27.94 (4.08) | 27.57 (3.84)
Time in dialysis [Mean (Standard Deviation); unit: months] | 37.86 (29.97) | 28.61 (23.61) | 32.95 (26.16) | 33.22 (26.82)
Glycated hemoglobin [Mean (Standard Deviation); unit: percentage] | 5.27 (0.51) | 5.37 (0.32) | 5.31 (0.43) | 5.31 (0.43)
Triglycerides levels [Mean (Standard Deviation); unit: mg/dl] | 184.26 (114.93) | 199.31 (91.99) | 209.69 (109.01) | 197.60 (105.83)
Total cholesterol [Mean (Standard Deviation); unit: mg/dl] | 165.86 (47.99) | 162.82 (39.29) | 179.37 (42.47) | 169.40 (43.78)
HDL-c [Mean (Standard Deviation); unit: mg/dl] | 40.95 (14.37) | 42.50 (12.07) | 42.21 (15.27) | 41.85 (13.92)
LDL-c [Mean (Standard Deviation); unit: mg/dl] | 98.45 (36.61) | 90.00 (37.53) | 103.81 (36.03) | 97.65 (36.79)
Fasting blood glucose level [Mean (Standard Deviation); unit: mg/dl] | 91.91 (13.16) | 97.74 (14.29) | 91.90 (13.93) | 93.85 (13.96)
Transfusions [Mean (Standard Deviation); unit: average number of transfusions/patient] | 0.66 (1.27) | 0.85 (2.50) | 0.83 (2.12) | 0.78 (1.99)
Cold ischemia time [Mean (Standard Deviation); unit: hours] | 16.83 (5.52) | 18.15 (5.40) | 17.26 (6.36) | 17.41 (5.75)
Age of the donor [Mean (Standard Deviation); unit: years] | 62.11 (10.43) | 62.88 (8.92) | 61.62 (10.02) | 62.20 (9.75)
Donor creatinine levels [Mean (Standard Deviation); unit: mg/dl] | 0.80 (0.28) | 0.83 (0.40) | 0.87 (0.29) | 0.83 (0.32)
Human leucocyte antigens (HLA) class I (A, B) and class II (DR) incompatibilities [Mean (Standard Deviation); unit: number of incompatibilities] | 3.55 (1.17) | 4.00 (0.87) | 4.24 (1.10) | 3.93 (1.10)
Anti-HLA lymphocytotoxic antibodies against <25% a reference panel [Number; unit: participants]
  Yes | 3 | 0 | 1 | 4
  No Antibodies | 41 | 40 | 40 | 121
  Not available | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure "New Onset Diabetes After Renal Transplantation" (NODAT)
Description: American Diabetes Association criteria (ADA) including an oral glucose tolerance test.
Time Frame: 1 year
Population: Participants analyzed: participants living with a functioning graft at study end
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 41 | 39 | 38
percentage of participants
  % of patients with NODAT | 34.1 [21.6 to 49.5] | 23.1 [12.7 to 38.3] | 7.9 [2.7 to 20.8]
  % of patients without NODAT | 65.9 [50.5 to 78.4] | 76.9 [61.6 to 87.3] | 92.1 [79.2 to 97.3]
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.02, Chi-squared

2. Primary Outcome: Patients Treated With Insulin or Oral Antidiabetic Drugs
Time Frame: 1 year
Population: Participant analyzed: participants living with a functioning graft at study end.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 41 | 39 | 38
percentage of participants | 20 [10.5 to 34.8] | 15.4 [7.3 to 29.7] | 2.6 [0.5 to 13.5]
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.06, Chi-squared

3. Primary Outcome: Primary Outcome Measure (Glucose Intolerance)
Description: Glycemia >=140 and <200 mg/dl, 2 hours after a standard oral glucose tolerance test. Measured values: glucose intolerance at 1 year defined by ADA criteria.
Time Frame: 1 year
Population: Participants included are those that did not develop NODAT based on not reporting the use of anti-diabetic drugs plus a fasting plasma glucose <126 mg/dl .
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 26 | 29 | 30
percentage of participants | 26.9 [13.7 to 46.1] | 31.0 [17.3 to 49.2] | 33.3 [19.2 to 51.2]
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.9, Chi-squared

4. Secondary Outcome: Rejection
Description: Biopsy proven acute rejection. Measured variable: Rate of Biopsy proven acute rejection.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 44 | 42 | 42
percentage of participants | 11.4 [4.95 to 24.0] | 4.8 [1.3 to 15.8] | 21.4 [11.7 to 36.0]
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.07, Chi-squared

5. Secondary Outcome: Renal Function
Description: Estimated Glomerular Filtration Rate (ml/min/1.73 m^2)
Time Frame: 1 year
Population: Participants analyzed: Participants living with a functioning graft at study end.
Measure: Mean (95% Confidence Interval); unit: ml/min/1.73 m^2
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 41 | 39 | 38
ml/min/1.73 m^2 | 51.9 [45.2 to 58.5] | 47.4 [42.9 to 52.0] | 44.6 [37.8 to 51.3]
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.2, ANOVA

6. Secondary Outcome: Proteinuria
Time Frame: 1 year
Population: Participants analyzed: participants living with a functioning graft at study end.
Measure: Mean (95% Confidence Interval); unit: mg/day
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 39 | 36 | 36
mg/day | 208 [121 to 296] | 241 [110 to 373] | 343.2 [154 to 532]
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.4, ANOVA

7. Secondary Outcome: Blood Pressure
Description: Systolic pressure (mmHg)
Time Frame: 1 year
Population: Participants analyzed: participants living with a functioning graft at study end.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 39 | 39 | 36
mmHg | 135.36 (15.75) | 133.97 (13.67) | 136.28 (17.27)
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.8, ANOVA

8. Secondary Outcome: Blood Pressure
Description: Diastolic pressure (mmHg)
Time Frame: 1 year
Population: Participants analyzed: participants living with a functioning graft at study end.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 39 | 39 | 36
mmHg | 76.67 (8.93) | 74.59 (9.83) | 76.64 (10.27)
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.56, ANOVA

9. Secondary Outcome: Number of Antihypertensive Drugs Patients Reported Taking.
Time Frame: 1 year
Population: Participants analyzed: participants living with a functioning graft at study end.
Measure: Median (Inter-Quartile Range); unit: number of antihypertensive drugs
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 41 | 39 | 38
number of antihypertensive drugs | 2 [1 to 3] | 2 [1 to 2] | 2 [1 to 2]
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.8, Kruskal-Wallis

10. Secondary Outcome: Lipidic Profile (Triglycerides)
Time Frame: 1 year
Population: Participants analyzed: participants living with a functioning graft at study end.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 39 | 37 | 37
mg/dl | 159.44 (93.68) | 145.59 (52.97) | 160.78 (84.26)
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.66, ANOVA

11. Secondary Outcome: Lipidic Profile (Cholesterol)
Description: Lipidic Profile (total cholesterol)
Time Frame: 1 year
Population: Participants analyzed: participants living with a functioning graft at study end.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 39 | 37 | 38
mg/dl | 169.05 (30.57) | 178.24 (33.64) | 168.89 (33.38)
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.37, ANOVA

12. Secondary Outcome: Lipidic Profile (HDL-c)
Time Frame: 1 year
Population: Participants analyzed: participants living with a functioning graft at study end.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 38 | 35 | 34
mg/dl | 44.84 (13.89) | 49.29 (16.90) | 48.35 (16.59)
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.45, ANOVA

13. Secondary Outcome: Lipidic Profile (LDL-c)
Time Frame: 1 year
Population: Participants analyzed: participants living with a functioning graft at study end.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 37 | 35 | 34
mg/dl | 94.00 (27.04) | 95.43 (26.54) | 88.65 (25.73)
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.50, ANOVA

14. Secondary Outcome: Percentage of Patients Using Statins
Time Frame: 1 year
Population: Participants analyzed: participants living with a functioning graft at study end.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 41 | 39 | 38
percentage of participants | 56. [41 to 70] | 61.5 [45.9 to 75.1] | 73.7 [58 to 85]
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.17, Chi-squared

15. Secondary Outcome: Changes of Carotid Intima-media Thickness Over Time
Description: absolute difference between carotid intima-media thickness at study end versus baseline.
Time Frame: 1 year
Population: Participants analyzed: participants living with a functioning graft at study end.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 9 | 8 | 10
mm | 0.12 [0.09 to 0.15] | 0.04 [-0.15 to 0.23] | 0.01 [-0.01 to 0.03]
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.5, ANOVA

16. Secondary Outcome: Percentage of Patients Using Acetylsalicylic Acid (ASA)
Time Frame: 1 year
Population: Analysis population description: participants living with a functioning graft at study end.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Number analyzed (Participants) | 39 | 37 | 36
percentage of participants | 53.9 [38.6 to 68.4] | 48.7 [33.5 to 64.1] | 52.8 [37 to 68]
Statistical Analysis 1: Comparison: Tacrolimus With Rapid Steroid Withdrawal vs Tacrolimus With Steroids Minimization vs CsA With Steroid Minimization; Test type: Superiority or Other; p = 0.9, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tacrolimus With Rapid Steroid Withdrawal | Tacrolimus With Steroids Minimization | CsA With Steroid Minimization
Serious Adverse Events (participants affected / at risk) | 8/44 | 5/42 | 12/42
Other Adverse Events (participants affected / at risk) | 12/44 | 17/42 | 18/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus With Rapid Steroid Withdrawal (N=44) | Tacrolimus With Steroids Minimization (N=42) | CsA With Steroid Minimization (N=42)
Heart attack resulting in death event (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Shock resulting in death event (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Rejection (Immune system disorders) | 5 (5) | 2 (2) | 9 (9)
Graft Loss (Immune system disorders) | 1 (1) | 2 (2) | 2 (2)
Pneumonia resulting in death event (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis resulting in death event (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus With Rapid Steroid Withdrawal (N=44) | Tacrolimus With Steroids Minimization (N=42) | CsA With Steroid Minimization (N=42)
Acute Miocardial Infarction or Coronary Revascularization (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Stroke (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
BK Virus Infection (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
CMV Infection (Infections and infestations) | 7 (7) | 6 (6) | 12 (12)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Acute Pyelonephritis of the graft (Infections and infestations) | 2 (2) | 6 (6) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 5 (5) | 1 (1)
Neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No